CLINICAL TRIAL: NCT06947681
Title: Factors Predicting and Assessment of Post Dialysis Fatigue in Patients on Regular Hemodialysis in Assiut University Hospital
Brief Title: we Use Recovery Time to Assess Post-dialysis Fatigue and we Use Also Two Different Fatigue Scales 1- Visual Analogue Scale 2- Fatigue Severity Scale and we Address Risk Factors of PDF and Apply the Scales on Regular Hemodialysis Patients in Hemodialysis Unit of Assiut University Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Christina Kamel Hanna Soliman, resident, Assiut University
Other Study IDs: post-dialysis fatigue
Record Dates: First submitted 2025-03-16; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-03

CONDITIONS: Post-dialysis Fatigue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- adult patients on regular hemodialysis on assiut university hospitals: no intervention

SUMMARY:
To improve the quality of life of hemodialysis patients and provide better control for post dialysis fatigue in regular hemodialysis patients.

DETAILED DESCRIPTION:
Post-dialysis fatigue (PDF) is a prevalent and debilitating symptom among patients undergoing regular hemodialysis, characterized by a persistent sense of physical and mental exhaustion following dialysis sessions This condition adversely affects patients' quality of life, daily functioning, and adherence to treatment regimens .Despite its high prevalence, PDF remains under-recognized and inadequately addressed in clinical practice. The etiology of PDF is multifactorial, encompassing physiological, psychological, and lifestyle-related factors. Recent studies have identified several predictors of PDF, including sleep disorders, the presence of comorbidities, the number of weekly dialysis sessions, and the duration of hemodialysis treatment . The symptoms and severity of PDF are evaluated using various scales. In cases of PDF, to examine the subjective symptoms of patients themselves, it is useful to utilize patient-based outcomes. However, in conventional PDF studies, the evaluation indices have not been uniform. First, in studies evaluating fatigue after dialysis based on the "time," "frequency," and "intensity" the reliability and validity of the scales were not examined. Second, the recovery time is not an index that measures PDF directly but instead an indirect indicator that measures the "time to recover from hemodialysis." Third, the fatigue scale does not measure true PDF but rather chronic fatigue experienced by dialysis patients .

in that research we use time recovery to assess post-dialysis fatigue and we use also two different fatigue scales visual analogue scale to evaluate fatigue severity and fatigue severity scale In that research we address risk factors of PDF and apply the scales on regular hemodialysis patients in hemodialysis unit of Assiut University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* • End stage renal diseases (ESRD) patients who receive hemodialysis 3 times a week for 4 h each time.

  * > 20 years of age.
  * Both sexes.
  * Patients with stable clinical examination.
  * Patients who receiving hemodialysis for more than 3 months.
  * All patients were able to go to the center for hemodialysis on their own.
  * All patients who accept to share in the research.

Exclusion Criteria:

* • Ages below 20 years.

  * Patients with severe cardiovascular and cerebrovascular diseases.
  * Mental illness that is difficult to diagnose and treat.
  * Surgery within the past month.
  * Patients with acute infections.
  * Pregnancy.
  * Presence of malignancy.
  * Undergoing fracture treatment, and serious mobility.
  * patients with eye problems.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients on regular hemodialysis on hemodialysis unit of assiut university hospital
Sampling Method: Non-Probability Sample
Enrollment: 155 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Identification of predictive factors significantly associated with post-dialysis fatigue | about 2 years
  Demographic, clinical, psychological factors significantly associated with post-dialysis fatigue.

SECONDARY OUTCOMES:
Determination of the most effective assessment tool for measuring post dialysis fatigue. | about 2 years
  assessment tool for measuring post dialysis fatigue by using recovery time recovery time of post dialysis is time to recover from hemodialysis
Estimated prevalence of post-dialysis fatigue in the study population. | about 2 years
  by using a questionnaire
Estimated severity of post-dialysis fatigue in the study population. | about 2 years
  by using questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: christina kamel hanaa, master degree, Principal Investigator — Assiut University; Hoida AbdAlhakam Nafady, professor, Study Director — Assiut University; Noha Gamal Abd Elmalek, doctor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided
it will be discussed with my supervisoirs

REFERENCES:
- [Background] Kodama, H., Togari, T., Konno, Y. et al. A new assessment scale for post-dialysis fatigue in hemodialysis patients. Ren Replace Ther 6, 1 (2020). https://doi.org/10.1186/s41100-019-0252-5
- [Background] Dou J, Liu H, Ma Y, Wu YY, Tao XB. Prevalence of post-dialysis fatigue: a systematic review and meta-analysis. BMJ Open. 2023 Jun 13;13(6):e064174. doi: 10.1136/bmjopen-2022-064174. PMID 37311633
- [Background] Sklar AH, Riesenberg LA, Silber AK, Ahmed W, Ali A. Postdialysis fatigue. Am J Kidney Dis. 1996 Nov;28(5):732-6. doi: 10.1016/s0272-6386(96)90256-5. PMID 9158212
- [Background] Faioli A, Bergesio G, Sama C, Gallo B. Predictors of Fatigue Among Patients on Hemodialysis: An Observational Study. Cureus. 2024 Aug 1;16(8):e65953. doi: 10.7759/cureus.65953. eCollection 2024 Aug. PMID 39221326
- See also: Website for a linked papers and articles — https://pubmed.ncbi.nlm.nih.gov/
- See also: Search engine that' includes research similar articles or papers — https://scholar.google.com/
- Available data/document: Study Protocol: Not available at moment — https://pubmed.ncbi.nlm.nih.gov/ — Most of the informations available at This site and Google Scholar